CLINICAL TRIAL: NCT03211065
Title: The Use of 20% Subcutaneous Immunoglobulin Replacement Therapy in Patients With B Cell Non Hodgkin's Lymphoma With Humoral Immune Dysfunction After Treatment With Rituximab
Brief Title: Humoral Immunodeficiency With Rituximab and Therapy With Subcutaneous Ig
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, S. Shahzad Mustafa, Physician, Associate Medical Director, Rochester General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT16-34083
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2020-08

CONDITIONS: Secondary Immune Deficiency
Keywords: Rituximab; Non Hodgkin's Lymphoma; Subcutaneous Immunoglobulin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Hizentra

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Immunoglobulin therapy (Experimental): Patients with abnormal humoral function following treatment with rituximab will be treated with 20% subcutaneous immunoglobulin.
  Interventions: Drug: 20% subcutaneous immunoglobulin

INTERVENTIONS:
Drug: 20% subcutaneous immunoglobulin — Subcutaneous Immunoglobulin
  Other Names: Cuvitru

SUMMARY:
To study the use of subcutaneous (injected under the skin) immunoglobulin replacement therapy (replacement of antibodies, which are infection-fighting proteins) in patients with a type of blood cancer called lymphoma, who have been treated with rituximab (a type of chemotherapy) and have an abnormal immune system putting them at increased risk of infection.

DETAILED DESCRIPTION:
The investigators propose evaluating patients with B cell non-Hodgkin's lymphoma treated with rituximab within the past 2 years with baseline immunoglobulin levels and vaccine responses to polysaccharide (pneumococcus, meningococcus) and peptide (tetanus, diphtheria) antigens. Patients with impaired vaccine responses may benefit most from immunoglobulin prophylaxis and will be proactively started on 20% subcutaneous replacement therapy. This study is novel in that it will stratify patients according to their humoral response to polysaccharide and peptide vaccines, and will proactively initiate therapy with the new 20% subcutaneous immunoglobulin in those with impaired humoral response rather than starting it after infections occur. This will potentially lead to decreased infections and improved quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of B cell non-Hodgkin's lymphoma
2. Medically stable
3. Able to understand and willingness to sign a written informed consent
4. Able to comply with study procedures

Exclusion Criteria:

1. Previously diagnosed primary immunodeficiency
2. Additional immunosuppressive states
3. Ongoing therapy with Ig replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Number of non-neutropenic infections per subject requiring antibiotics in the year after enrollment | 1 year
  How many antibiotics are prescribed in one year for any type of infection

SECONDARY OUTCOMES:
Quality of life score for participants during the one year enrollment | 1 year
  Assessed with Short Form 36 (SF 36)

CONTACTS AND LOCATIONS:
Overall Officials: S Shahzad Mustafa, MD, Principal Investigator — Rochester Regional Health
Locations (1):
- Allergy and Immunology, 222 Alexander Street, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan B, Kopyltsova Y, Khokhar A, Lam F, Bonagura V. Rituximab and immune deficiency: case series and review of the literature. J Allergy Clin Immunol Pract. 2014 Sep-Oct;2(5):594-600. doi: 10.1016/j.jaip.2014.06.003. Epub 2014 Aug 7. PMID 25213054
- [Background] Davis TA, White CA, Grillo-Lopez AJ, Velasquez WS, Link B, Maloney DG, Dillman RO, Williams ME, Mohrbacher A, Weaver R, Dowden S, Levy R. Single-agent monoclonal antibody efficacy in bulky non-Hodgkin's lymphoma: results of a phase II trial of rituximab. J Clin Oncol. 1999 Jun;17(6):1851-7. doi: 10.1200/JCO.1999.17.6.1851. PMID 10561225
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- [Background] Kimby E. Tolerability and safety of rituximab (MabThera). Cancer Treat Rev. 2005 Oct;31(6):456-73. doi: 10.1016/j.ctrv.2005.05.007. Epub 2005 Jul 28. PMID 16054760
- [Background] Kelesidis T, Daikos G, Boumpas D, Tsiodras S. Does rituximab increase the incidence of infectious complications? A narrative review. Int J Infect Dis. 2011 Jan;15(1):e2-16. doi: 10.1016/j.ijid.2010.03.025. Epub 2010 Nov 11. PMID 21074471
- [Background] van Oers MH, Klasa R, Marcus RE, Wolf M, Kimby E, Gascoyne RD, Jack A, Van't Veer M, Vranovsky A, Holte H, van Glabbeke M, Teodorovic I, Rozewicz C, Hagenbeek A. Rituximab maintenance improves clinical outcome of relapsed/resistant follicular non-Hodgkin lymphoma in patients both with and without rituximab during induction: results of a prospective randomized phase 3 intergroup trial. Blood. 2006 Nov 15;108(10):3295-301. doi: 10.1182/blood-2006-05-021113. Epub 2006 Jul 27. PMID 16873669
- [Background] Casulo C, Maragulia J, Zelenetz AD. Incidence of hypogammaglobulinemia in patients receiving rituximab and the use of intravenous immunoglobulin for recurrent infections. Clin Lymphoma Myeloma Leuk. 2013 Apr;13(2):106-11. doi: 10.1016/j.clml.2012.11.011. Epub 2012 Dec 29. PMID 23276889
- [Background] Cabanillas F, Liboy I, Pavia O, Rivera E. High incidence of non-neutropenic infections induced by rituximab plus fludarabine and associated with hypogammaglobulinemia: a frequently unrecognized and easily treatable complication. Ann Oncol. 2006 Sep;17(9):1424-7. doi: 10.1093/annonc/mdl141. PMID 16966368
- [Background] Duraisingham SS, Buckland M, Dempster J, Lorenzo L, Grigoriadou S, Longhurst HJ. Primary vs. secondary antibody deficiency: clinical features and infection outcomes of immunoglobulin replacement. PLoS One. 2014 Jun 27;9(6):e100324. doi: 10.1371/journal.pone.0100324. eCollection 2014. PMID 24971644
- [Background] Makatsori M, Kiani-Alikhan S, Manson AL, Verma N, Leandro M, Gurugama NP, Longhurst HJ, Grigoriadou S, Buckland M, Kanfer E, Hanson S, Ibrahim MA, Grimbacher B, Chee R, Seneviratne SL. Hypogammaglobulinaemia after rituximab treatment-incidence and outcomes. QJM. 2014 Oct;107(10):821-8. doi: 10.1093/qjmed/hcu094. Epub 2014 Apr 28. PMID 24778295
- [Background] Spadaro G, Pecoraro A, De Renzo A, Della Pepa R, Genovese A. Intravenous versus subcutaneous immunoglobulin replacement in secondary hypogammaglobulinemia. Clin Immunol. 2016 May;166-167:103-4. doi: 10.1016/j.clim.2016.04.001. Epub 2016 Apr 7. PMID 27063866
- [Background] Compagno N, Cinetto F, Semenzato G, Agostini C. Subcutaneous immunoglobulin in lymphoproliferative disorders and rituximab-related secondary hypogammaglobulinemia: a single-center experience in 61 patients. Haematologica. 2014 Jun;99(6):1101-6. doi: 10.3324/haematol.2013.101261. Epub 2014 Mar 28. PMID 24682509
- [Background] Cooper N, Arnold DM. The effect of rituximab on humoral and cell mediated immunity and infection in the treatment of autoimmune diseases. Br J Haematol. 2010 Apr;149(1):3-13. doi: 10.1111/j.1365-2141.2010.08076.x. Epub 2010 Feb 11. PMID 20151975